CLINICAL TRIAL: NCT05886816
Title: Mitoquinone/mitoquinol Mesylate As Oral and Safe Postexposure Prophylaxis for Covid-19
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Theodoros Kelesidis, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB#STU-2023-0524
Record Dates: First submitted 2023-06-01; First posted 2023-06-02 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: SARS-CoV Infection; COVID-19
Keywords: SARS-CoV Infection; COVID-19; Post-exposure prophylaxis
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19 | interventions — mitoquinone

STUDY DESIGN:
Intervention Model Description: Group 1: Mito-MES 20 mg daily initiated within 3 days post exposure and taken daily during the study Group 2: Placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study participants and the investigators involved in the acquisition and analysis of key outcomes will be blinded to the group status of the subjects. The double-blind drugs will be labelled within the institutional investigational drug service pharmacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mito-MES (Experimental): MitoQ pills 20 mg orally daily taken during the study and initiated within 3 days post exposure.
  Interventions: Drug: Mitoquinone/mitoquinol mesylate
- Control group (Placebo Comparator): Placebo pills orally daily taken during the study and initiated within 3 days post exposure.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mitoquinone/mitoquinol mesylate — Mitochondrial antioxidant
  Arms: Mito-MES
Other: Placebo — Placebo pills
  Arms: Control group

SUMMARY:
Adults who do not have major health, kidney, gastrointestinal disease will be randomized to receive oral mitoquinone/mitoquinol mesylate (Mito-MES) versus placebo to prevent the development and progression of COVID-19 after high-risk exposure to a person with confirmed SARS-CoV-2 infection.

DETAILED DESCRIPTION:
The overall goal of the study is to determine the efficacy of the treatment with mito-MES 20 mg daily versus placebo for 14 days to prevent confirmed SARS-CoV-2 infection in high-risk close contacts of confirmed COVID-19 cases. Primary measure will be confirmed COVID-19 infection based on a diagnostic test within 14 days after exposure. Secondary measures of efficacy will be symptomatic viral infection, hospitalization, respiratory failure requiring ventilatory support attributable to COVID-19 disease, mortality. The secondary objective is to determine the safety of mito-MES for 14 days as post-exposure prophylaxis against SARS-CoV-2 in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

Age 18-65 years old Asymptomatic (no symptoms of viral infection) on study entry High risk exposure without use of masks to confirmed case of COVID-19 Members in a household one of which is a confirmed case of COVID-19 Negative baseline SARS-COV-2 diagnostic test

Exclusion Criteria:

* Women with variations in physiological functions due to hormones that may effect immune function and (transgender, pregnant, breastfeeding)
* Specific significant clinical diseases [cardiovascular disease (such as coronary artery/vascular disease), heart disease (such as congestive heart failure, cardiomyopathy, atrial fibrillation), lung disease (such as chronic obstructive pulmonary disease, asthma, bronchiectasis, pulmonary fibrosis, pleural effusions), kidney disease (glomerular filtration rate or GFR less than 60 ml/min/1.73 m2), liver disease (such as cirrhosis, hepatitis), major immunosuppression (such as history of transplantation, uncontrolled HIV infection, cancer on active chemotherapy] based on history. Participants with well controlled HIV (CD4 count > 500 cells/mm^3 and HIV viral load < 50 copies/ml) and people with remote history of cancer not on active treatment will be allowed to participate.
* History of known gastrointestinal disease (such as gastroparesis) that may predispose patients to nausea
* History of auto-immune diseases
* Chronic viral hepatitis
* Use of systemic immunomodulatory medications (e.g. steroids) within 4 weeks of enrollment
* Any participant who has received any investigational drug within 30 days of dosing
* History of underlying cardiac arrhythmia
* History of severe recent cardiac or pulmonary event
* A history of a hypersensitivity reaction to any components of the study drug or structurally similar compounds including Coenzyme Q10 and idebenone
* Unable to swallow tablets
* Use of any investigational products within 4 weeks of enrollment
* Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study requirements.
* Eligible for other FDA approved treatment for post-exposure prophylaxis against SARS-CoV-2
* Use of Coenzyme Q10 or Vitamin E < 120 days from enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 infection | Within 14 days after exposure to SARS-CoV-2
  Confirmed SARS-CoV-2 infection based on a diagnostic test

SECONDARY OUTCOMES:
Safety of mito-MES | Within 14 days since initiation of the pills
  Side effects observed during use of mito-MES
Symptomatic SARS-CoV-2 infection | Within 14 days after exposure to SARS-CoV-2
  Development of symptomatic SARS-CoV-2 infection
Severity of symptoms of SARS-CoV-2 infection | Within 14 days after exposure to SARS-CoV-2
  Assessment of severity of symptoms of SARS-CoV-2 infection
Duration of symptoms of SARS-CoV-2 infection | Within 14 days after exposure to SARS-CoV-2
  Assessment of duration of symptoms of SARS-CoV-2 infection

CONTACTS AND LOCATIONS:
Overall Officials: Theodoros Kelesidis, MD, PHD, Msc, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No